CLINICAL TRIAL: NCT03210480
Title: Clinical Evaluation of Switching to Lithiofor® (Lithium Sulphate Slow -Release, Li-SR Tablets) From Carbolithium® (Lithium Carbonate Immediate-Release, Li-IR, Capsules) in Bipolar Patients, Poorly Tolerant to Lithium Immediate-release Treatment.
Brief Title: SALT Study (Switching to the Administration of Lithium Slow -Release Treatment)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor's decision due to slow enrollment rate.
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 136PO15274; 2016-001714-14 (EudraCT Number)
Record Dates: First submitted 2017-06-23; First posted 2017-07-07 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Disorder
Keywords: Lithium Sulphate; Prolonged release formulation; Lithium carbonate; Immediate release formulation; Bipolar Disorder; Tremor
MeSH Terms: conditions — Bipolar Disorder; Tremor

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Lithium sulphate prolonged-release 660 mg
  Interventions: Drug: Lithium sulphate prolonged-release 660 mg
- Group 2 (Active Comparator): Lithium carbonate immediate-release 150 mg and 300 mg
  Interventions: Drug: Lithium carbonate immediate-release 150 mg and 300 mg

INTERVENTIONS:
Drug: Lithium sulphate prolonged-release 660 mg — Oral administration of one tablet once or twice daily (one tablet in the morning and one tablet in the evening) or two tablets in a single dose (two tablets in the evening) of Lithium sulphate 660 mg (Lithium sulphate dose will be individualised for each patient according to the relevant SmPC). Treatment duration: 3 months.
  Other Names: LITHIOFOR®
  Arms: Group 1
Drug: Lithium carbonate immediate-release 150 mg and 300 mg — Oral administration of 300-1800 mg daily divided into 2-6 doses of Lithium carbonate capsules (Lithium carbonate dose will be individualised for each patient according to the relevant SmPC). Treatment duration: 3 months.
  Other Names: CARBOLITHIUM®
  Arms: Group 2

SUMMARY:
The aim of the study is to assess the tolerability, efficacy and safety of a new lithium sulphate prolonged release formulation (Lithiofor®) in patients affected by Bipolar Disorder poor tolerant to lithium immediate-release treatment in terms of lithium-induced tremor when switched from therapy with a lithium carbonate immediate release formulation (Carbolithium®) to a new lithium sulphate prolonged release formulation (Lithiofor®).

DETAILED DESCRIPTION:
This is a phase IV, randomized, open, parallel groups, multicentre, prospective study.

The main purpose of this clinical trial is to evaluate the change in the lithium induced tremor when switching from Lithium Immediate Release formulation (Carbolithium®) to Lithium Sulphate prolonged-release formulation (Lithiofor®) in Bipolar Disorder patients, poorly tolerant to the Lithium Immediate Release treatment. The primary end point will be the reduction of the lithium induced tremor.

Patients in treatment with lithium carbonate immediate-release (Carbolithium®), will be enrolled in the study and, after 1 week of maintaining treatment, will be randomly switched to Lithium prolonged-release formulation or will continue the previous therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years (limits included), with no limitation of race. Female patients with childbearing potential should have a negative pregnancy test and should not be breastfeeding. Male and female patients should use an appropriate birth control method.
2. Diagnosis of Bipolar disorder (BD) I or II (as per DSM-5), with or without rapid cycling.
3. BD patients in treatment with lithium Carbolithium® immediate-release, presenting at the screening and baseline low tolerability in terms of tremor (tremor severity assessment ≥ 2 on single item of the UKU side-effect rating scale).
4. MADRS score ≤ 10 and YMRS ≤ 12 at screening and baseline visits.
5. Patients legally capable to give the consent to participate in the study and available to sign and date the written informed consent.
6. Patient able to understand the study procedures and to comply with protocol requirements.

Exclusion Criteria:

1. Fulfilling criteria for the following disorders: schizophrenia, psychotic and schizoaffective disorders, unipolar depression; concomitant organic mental disorder or intellectual disability; history of dementia or cognitive disorders, any neurodegenerative diseases.
2. Known hypersensitivity or allergy to lithium or to any components of the study medications.
3. Pharmacological treatments affecting tremor, except for patients treated for at least 2 months before the screening visit (i.e. Beta-blockers; for further details).
4. Known tremor due to irreversible lithium neurotoxicity.
5. Patients at risk for suicidal behaviour.
6. Immunocompromised patients.
7. Acute, or chronic, or recurrent medical conditions that might affect/jeopardize the study results.
8. Significant liver disease, defined as known active hepatitis or elevated liver enzymes > 3 times the upper boundary of the normal ranges.
9. Value of creatinine outside the normal ranges and judged clinically relevant by Investigator.
10. Any contraindication listed in the Summaries of Product Characteristics (SmPC) of Carbolithium® and lithium sulphate prolonged-release tablets (Lithiofor®).
11. Positive history for drugs.
12. Alcohol abuse.
13. Positive urine drug screen for CNS-active drugs (cocaine, opioids, amphetamines and cannabinoids) at Visit 0 (screening).
14. Clinically significant abnormalities on physical examination, vital signs, ECG, laboratory tests prior to screening visit.
15. Inability to comply with the protocol requirements, instructions and study-related restrictions; e.g. uncooperative attitude, inability to return for study-visits, and improbability of completing the clinical study.
16. Vulnerable subjects (e.g. persons kept in detention).
17. Participation to an interventional clinical study within 3 months prior to the screening visit.
18. If Subject is the Investigator or his(her) deputies, first grade relative, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Change of item 2.5 (tremor) in Udvalg for Kliniske Undersøgelser (UKU) scale | Baseline - Week 1
  Proportion of patients with an improvement in tremor assessed by the change from baseline of item 2.5 in UKU side-effect rating scale after 1-week treatment period.

SECONDARY OUTCOMES:
Change of item 2.5 (tremor) in Udvalg for Kliniske Undersøgelser (UKU) scale | Baseline - Weeks 4 and 12
  Proportion of patients with an improvement in tremor assessed by the change from baseline of item 2.5 in UKU side-effect rating scale after 4- and 12-week treatment period.
Change of item 3.8 in Udvalg for Kliniske Undersøgelser (UKU) scale | Baseline - Weeks 1, 4 and 12
  Proportion of patients with a change from baseline of item 3.8 in UKU side-effect rating scale after 1-, 4- and 12-week treatment period.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline - Weeks 1, 4 and 12
  Change from baseline of total score in MADRS scale after 1-, 4- and 12-week treatment period.
Change in Young Mania Rating Scale (YMRS) | Baseline - Weeks 1, 4 and 12
  Change from baseline of total score in YMRS scale after 1-, 4- and 12-week treatment period.
Change in Treatment Satisfaction Questionnaire for Medication (TSQM) scale | Baseline - Weeks 1 and 12
  Change from baseline in each sub-scale of TSQM after 1- and 12-week treatment period.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) | Baseline - Weeks 1 and 12
  Change from baseline in Q-LES-Q-SF after 1- and 12-week treatment period.
Change in Clinical Global Impression (CGI) scale | Baseline - Weeks 1 and 12
  Assessment by the physician of the overall efficacy by CGI scale after 1- and 12-week treatment period.
Frequency of treatment-related adverse events | 12 weeks
  Monitoring of the frequency of adverse events, physical examination, vital signs, ECG, laboratory analyses, plasma Lithium concentration.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Ospedale San Giovanni di Dio di Orbetello Unità Funzionale Salute Mentale, Orbetello, Grosseto
  - Azienda Ospedaliera Papa Giovanni XXIII - Servizio Psichiatrico di Diagnosi e Cura (SPDC 1), Bergamo
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST - Clinica Psichiatrica, Genova
  - Azienda Ospedaliera Universitaria Pisana - Psichiatria 1, Pisa
  - Azienda Ospedaliera Sant'Andrea - Dip. Di Neuroscienze, Salute mentale e Organi di senso- NESMOS, Roma
  - Azienda Ospedaliera Universitaria Senese - Dip. Interaziendale di salute mentale - Psichiatria, Siena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.angelinipharma.com